CLINICAL TRIAL: NCT05564728
Title: A Feasibility Study of a Conversational Agent App for Empowering Foot Care Literacy Among People With Diabetes and Their Carers
Brief Title: Diabetes Footcare Companion App for Patients and Carers
Status: Completed | Type: Observational
Sponsor: Nanyang Technological University (Other)
Collaborators: Tan Tock Seng Hospital (Other); Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Ho Hau Yan Andy, Joint Associate Professor, Lee Kong Chian School of Medicine, Nanyang Technological University
Other Study IDs: NanyangTU_WellFeet
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus Foot Ulcer; Diabetes Mellitus, Type 2; Diabetic Foot; Diabetic Foot Infection; Ulcer Foot; Ulcer, Leg
Keywords: Conversational Agent; Chatbot; Diabetes Literacy; Diabetes Knowledge; Self Management; Digital Therapeutics; Digital Health
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2; Foot Ulcer; Leg Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: All participants will receive a conversational agent app, Well Feet, to support them in learning foot care self-management.
  Interventions: Other: Conversational Agent/Chatbot App

INTERVENTIONS:
Other: Conversational Agent/Chatbot App — Well Feet is developed based on adaptive learning frameworks to deliver diabetes foot care education through a conversational agent. The learning path for each participant will be customised based on their responses to pre-module quizzes.
  Other Names: Well Feet

SUMMARY:
Diabetes education and self-management support can be delivered via mobile phones. This protocol aims to assess the feasibility and acceptability of Well Feet, a conversational agent, as a diabetic foot care companion. By utilizing feedback and responses to evaluative questions posted on the app's interface, the investigators intend to examine the app's technical, functional, and operational feasibility.

DETAILED DESCRIPTION:
Diabetes puts patients with diabetes at risk of foot complications. Besides well managed diabetes, providing diabetes foot care education and self-management support is key to reducing the risk of developing diabetic foot ulcers, a serious and costly complication of diabetes. Although, education and self-management support for people with diabetes can improve patients' quality of life, they are still commonly not provided or inadequate. Digital technologies have the potential to offer a new convenient, interactive, and engaging mode of self-management education and support.

This study aims to examine the feasibility of the Well Feet app for diabetes foot care education and self-management support in promoting optimal foot care behaviour. In recognizing that many people with diabetes, especially the elderly, require the support of informal carers, the app also targets their knowledge and support needs.

ELIGIBILITY:
Inclusion criteria for patients:

1. Patients diagnosed with type 2 diabetes and attending Tan Tock Seng Hospital Diabetes Clinic
2. Aged 21 years or above
3. Able to speak and read English
4. Own a smartphone or tablet
5. Can download the app
6. Have internet access
7. Able to give informed consent
8. Singapore nationality or permanent residents

Inclusion criteria for carers:

1. Provide care for a type 2 diabetes patient for the past 6 months
2. Aged 21 years or above
3. Able to speak and read English
4. Own a smartphone or tablet
5. Can download the app
6. Have internet access
7. Able to give informed consent

Exclusion criteria for patients and carers:

1. Pregnant
2. Inpatient
3. Received formal training in medicine or allied health services

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with type 2 diabetes and their carer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Usability of a health app among patients and carers at the end of the trial (1 month) | end-of-trial (1 month)
  A validated questionnaire, MHealth App Usability Questionnaire, will be used to determine the usefulness and applicability of an app with a conversational agent/chatbot among patients and carers. The questionnaire consists of 3 subscales, which are ease of use (5 items), interface and satisfaction (7 items), and usefulness (6 items). Participants rate each of the items using a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The usability of the app is determined by the total and average of all statements-the higher the overall average, the better the usability of the app. However, if the average score is lower than 4, it means that the usability of the app is not good
Qualitative perspective on a conversational agent/chatbot app usage experience among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  A focus group discussion among the app user will be done to collect feedback on the user experience at the end of the trial. Qualitative data on app usability, app applicability, app relevance and user feedback will be retrieved from the focus group discussion.

SECONDARY OUTCOMES:
Changes in foot care knowledge among patients and carers at baseline and end-of-trial (1 month). | baseline and end-of-trial (1 month)
  A validated questionnaire, Foot Care Knowledge Questionnaire (FTC) will be used to evaluate changes in patient's and carer's knowledge on foot care from baseline to the end-of-trial. The questionnaire consists of 12 items to be rate true or false and the score will be presented in term of percentage of correct answer. Higher percentage of correct answers means higher level of foot care knowledge.
Changes in foot care related self-management behaviour among patients at baseline and end-of-trial (1 month). | baseline and end-of-trial (1 month)
  A validated questionnaire, Nottingham Assessment of Functional Footcare (Revised 2015) will be used to assess changes in patient's level of foot care related self-management behaviour from baseline to the end-of-trial. This questionnaire consists of 29 items on a 5-point Likert scale. The total number of scores will be added up and multiply the score by 1.115 to obtain the final score. Higher score means better self-management care.
Changes in carer's quality of life at the baseline and end-of-trial. | baseline and end-of-trial (1 month)
  A validated questionnaire, Brief Assessment Scale for Caregivers (BASC) will be used to determine changes in carer's quality of life and level of burden from caring for a person with diabetes. This questionnaire consists of 14 items clustered into 5 factors. The mean BASC score is computed by summing up the non-NA items in each factor, then dividing by the number of items that were not missing. This gave a score scaled from 0 to 3, with a higher score indicating better caregiver outcomes.
Login frequency in the conversational agent/chatbot app among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  Data on login frequency will be retrieved from the backend of the app at the end of trial.
Time spent on the app in the conversational agent/chatbot app among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  Data on total number of minutes spent on the app will be retrieved from the backend of the app at the end of trial.
Number of module accessed in the conversational agent/chatbot app among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  Data on total number of education module accessed will be retrieved from the backend of the app at the end of trial.
Number of module completed in the conversational agent/chatbot app among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  Data on number of education module completed will be retrieved from the backend of the app at the end of trial.
Module quizzes scores in the conversational agent/chatbot app among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  At the end of each module, users will be directed to a module quiz. Data on total scores for the module quizzes will be collected from the backend of the app at the end of trial.
Module rating in the conversational agent/chatbot app among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  At the end of each module, users will be prompted to rate their learning experience using a 5-point Likert scale. Data of the ratings on each of the modules will be collected from the backend of the app at the end of trial.
Overall app rating for the conversational agent/chatbot app among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  Upon completion of all learning modules, users will be prompted to rate their overall experience of using the app using a 5-point Likert scale. Data of the overall experience of app rating will be retrieved from the backend of the app at the end of trial.
Usability of a conversational agent/chatbot among patients and carers at the end of the trial (1 month). | end-of-trial (1 month)
  A validated questionnaire, Chatbot Usability Questionnaire, will be used to determine the usefulness and applicability of a conversational agent/chatbot among patients and carers at the end of the trial. This questionnaire consists of 16 items on a 5-point Likert scale. The mean score will be calculated using CUQ calculator available on the Ulster University website. This higher mean score means better chatbot usability.

CONTACTS AND LOCATIONS:
Overall Officials: Liew Hui Ling, MBBS, Principal Investigator — Tan Tock Seng Hospital
Locations (2):
- Singapore (2):
  - Nanyang Technological University, Center for Population Health Sciences, Lee Kong Chian School of Medicine, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Patient data will be anonymised and aggregated for analysis.

REFERENCES:
- [Background] Liew H, Pienkowska A, Ang CS, Mahadzir MDA, Goh KFI, Lodh N, Bojic I, Lawate A, Ong QC, Venkataraman K, Car J, Ho AHY. Empowering Foot Care Literacy Among People Living With Diabetes and Their Carers With an mHealth App: Protocol for a Feasibility Study. JMIR Res Protoc. 2023 Nov 21;12:e52036. doi: 10.2196/52036. PMID 37988150
- [Derived] Still CH, Harwell C, Killion C, Sattar A, Viswanath SE. OPtimizing Technology to Improve Medication Adherence and BP Control (OPTIMA-BP) Invention Versus Waitlisted Group in African American Adults with Hypertension: A Randomized Control Trial Protocol. Nursing (Auckl). 2025;15:29-41. doi: 10.2147/nrr.s491609. Epub 2025 Mar 24. PMID 40342512